CLINICAL TRIAL: NCT01203579
Title: Different Strategies Using Autoantibodies and/or CT in the Detection of Lung Cancer
Brief Title: Chest Computed Tomography (CT) Screening Study With Antibody Testing
Status: Withdrawn | Type: Observational
Why Stopped: Due to lack of funding
Sponsor: Mayo Clinic (Other)
Responsible Party: David Midthun, MD, Mayo Clinic
Other Study IDs: 10-003048
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Lung Cancer
Keywords: CDT-Lung,CT scan,lung cancer detection
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the value of EarlyCDT-Lung test and CT scan both in lung cancer detection and potential health economic outcomes.

DETAILED DESCRIPTION:
EarlyCDT-Lung test and CT scan both for lung cancer detection and potential economic outcomes.

ELIGIBILITY:
* Persons 50-75
* Asymptomatic for lung cancer
* Current or former (stopped smoking less than 10 years ago) cigarette smokers
* History of cigarette smoking of at least 20 pack years
* History of cigarette smoking with a family history of lung cancer which gives an individual a personal risk similar to a smoking history of 20 pk/years (i.e. 1% at 5 years).
* Mentally competent individuals to sign an informed consent.
* Healthy enough to undergo pulmonary resection or stereotactic body radiotherapy.
* A fully informed signed consent form must have been obtained.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Current or Former Smokers with >20 pack year history and or family history of lung cancer. Ages 50-75 years old
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Midthun, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States